CLINICAL TRIAL: NCT00810550
Title: Carotid Ultrasound in the Evaluation of Heart Failure
Acronym: CUE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Harmony R. Reynolds, MD, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCC CUE-HF
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease; Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LV systolic dysfunction (Other): Diagnostic Testing
  Interventions: Other: Carotid ultrasound

INTERVENTIONS:
Other: Carotid ultrasound — Measurement of intima-media thickness

SUMMARY:
Coronary artery disease (CAD, cholesterol plaque buildup in the heart arteries) is the most common cause of left ventricular systolic dysfunction (weakening of the heart muscle). The standard test to find coronary artery disease is coronary angiography. This test is highly accurate but is invasive and carries a small risk of complications. This study investigates ultrasound of the carotid (neck) arteries as a screening test for severe coronary artery disease as a cause of left ventricular systolic dysfunction. It is hypothesized that carotid ultrasound will have excellent negative predictive value for severe CAD.

DETAILED DESCRIPTION:
Coronary artery disease (CAD, cholesterol plaque buildup in the heart arteries) is the most common cause of left ventricular systolic dysfunction (weakening of the heart muscle). The standard test to find coronary artery disease is coronary angiography. This test is highly accurate but is invasive and carries a small risk of complications. This study investigates ultrasound of the carotid (neck) arteries as a screening test for severe coronary artery disease as a cause of left ventricular systolic dysfunction. It is hypothesized that carotid ultrasound will have excellent negative predictive value for severe CAD.

ELIGIBILITY:
Inclusion Criteria:

* LVEF 40% or less

Exclusion Criteria:

* Prior diagnosis of coronary or carotid obstructive atherosclerosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for severe CAD | 1 Day

SECONDARY OUTCOMES:
Diagnostic accuracy for significant CAD | 1 Day

REFERENCES:
- [Derived] Reynolds HR, Steckman DA, Tunick PA, Kronzon I, Lobach I, Rosenzweig BP. Normal intima-media thickness on carotid ultrasound reliably excludes an ischemic cause of cardiomyopathy. Am Heart J. 2010 Jun;159(6):1059-66. doi: 10.1016/j.ahj.2010.03.026. PMID 20569720